CLINICAL TRIAL: NCT06221163
Title: Sociological Study of the Life Courses of Young TRANSgender Patients Consulting the REProduction Medicine Department
Brief Title: Sociological Study of the Life Courses of Young TRANSgender Patients
Acronym: ParTransRep
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Mikael AGOPIANTZ, MCU-PH - ART Center coordinator, Central Hospital, Nancy, France
Other Study IDs: 2023PI015
Record Dates: First submitted 2023-04-06; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Transgenderism
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young transgender: Transgender patients consulting the Reproductive Medicine Department for a request related to the preservation of their fertility or hormone therapy, as well as parents/family members present at the time of the appointment.
  The ceiling is 20 interviews and 80 hours.
  Interventions: Other: collection of biographical and sociological data

INTERVENTIONS:
Other: collection of biographical and sociological data — collection of biographical and sociological data. Conducting non-directive interviews (life stories) with transgender patients consulting the Reproductive Medicine Department and their volunteer relatives. Patients are given a 'flyer' at the time of their consultation on which the interviewer's contact details are given. They are free to contact the interviewer to find out when and where an interview might take place (outside hospital).

SUMMARY:
The number of people consulting for a request related to trans identity is increasing sharply. The study monocentric qualitative study of discursive material aims to describe the diversity of practices and discourses mobilized by the people concerned and their relatives in the wake of work already carried out in the human sciences. Conducting non-directive interviews (life stories) with transgender patients consulting the Reproductive Medicine Department and their volunteer relatives.The ceiling is 20 interviews and 80 hours of observation.

DETAILED DESCRIPTION:
The number of people consulting for a request related to trans identity is increasing sharply. The study aims to describe the diversity of practices and discourses mobilized by the people concerned and their relatives in the wake of work already carried out in the human sciences.

The care pathway is a central determinant of transgender experiences and differentiated care pathways indicate differentiated relationships to medicalisation and gender, which translate into practices. For the moment, transgender people who do not wish to preserve their fertility or who are not hormonally treated are over-represented in the sample. It is extremely important to gain access to the population that turns to the Reproductive Medicine Service.

The consultation is a place where knowledge (medical, activist, etc.) circulates and meets, which can then be re-appropriated or negotiated by transgender people. While interviews alone are not enough to describe this re-appropriation and negotiation, it is possible to do so through observations of consultations.

Conducting non-directive interviews (life stories) with transgender patients consulting the Reproductive Medicine Department and their volunteer relatives.

The ceiling is 20 interviews and 80 hours of observation.

Patients are given a 'flyer' at the time of their consultation on which the interviewer's contact details are given. They are free to contact the interviewer to find out when and where an interview might take place (outside hospital).

The ceiling is 20 interviews and 80 hours of observation. Discussions during the interview are recorded using a voice recording device, then transcribed in full in Word and anonymised. Discussions during consultations were recorded using notes, then formatted in Word and anonymised.

ELIGIBILITY:
Inclusion Criteria:

* transgender

Exclusion Criteria:

* Refusal by the patient.
* Refusal by the patient's legal guardian.
* Person under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender will be included. Male and female, non binary.
Study Population: Young transgender people
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Ethnographic observations of consultations to study relation to care pathway for transgender people | 1 year
  Conducting non-directive interviews (life stories) with transgender patients consulting the Reproductive Medicine Department and their volunteer relatives. Patients are given a flyer at the time of their consultation on which the interviewer's contact details are given. They are free to contact the interviewer to find out when and where an interview might take place (outside hospital).

SECONDARY OUTCOMES:
Ethnographic observations of transgender consultations in the Reproductive Medicine Department | 1 year
  Ethnographic observations of consultations in the Reproductive Medicine Department. The investigator is present during consultations with transgender patients and takes notes of what he observes and hears. He ensures that those present give their informed consent at the start of the appointment.

IPD SHARING:
Plan to Share IPD: No